CLINICAL TRIAL: NCT02770196
Title: Farm Fresh Foods for Healthy Kids: Innovative Community Supported Agriculture Cost-Offset Intervention to Prevent Childhood Obesity and Strengthen Local Agricultural Economies
Brief Title: Intervention Study of Cost-Offset Community Supported Agriculture (CO-CSA)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cornell University (Other)
Collaborators: University of Vermont (Other); University of North Carolina, Chapel Hill (Other); The Evergreen State College (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB #: 1501005266; 2015-68001-23230 (Other Grant/Funding Number: NIFA, USDA)
Record Dates: First submitted 2016-04-05; First posted 2016-05-12 (Estimated); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Pediatric Obesity; Child Nutrition Disorders
Keywords: Community-Supported Agriculture; Local Food System; Vegetable; Fruit; Childhood Obesity
MeSH Terms: conditions — Pediatric Obesity; Child Nutrition Disorders | interventions — Nutrition Assessment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group One (Two-year Intervention, 2016 Enrollment) (Experimental): Group one intervention participants in CO-CSA plus nutrition education will receive a subsidized share of CSA produce (50% standard member price) weekly for approximately 20 weeks each year in 2016 and 2017. During the 2016 season they will attend nine skill-based, nutrition education sessions focused on use of CSA produce.
  Interventions: Behavioral: CO-CSA plus Nutrition Education
- Group Two (Delayed Two-year Intervention, 2016 Enrollment) (Experimental): Group two intervention participants in CO-CSA plus nutrition education will receive a subsidized share of CSA produce (50% standard member price) weekly for approximately 20 weeks each year in 2017 and 2018. During the 2017 season they will attend nine skill-based, nutrition education sessions focused on use of CSA produce.
  Interventions: Behavioral: CO-CSA plus Nutrition Education
- Group Three (One-year Intervention, 2017 Enrollment) (Experimental): Group three intervention participants in CO-CSA plus nutrition education will receive a subsidized share of CSA produce (50% standard member price) weekly for approximately 20 weeks in 2017 and will attend nine skill-based, nutrition education sessions focused on use of CSA produce.
  Interventions: Behavioral: CO-CSA plus Nutrition Education
- Group Four (Delayed One-year Intervention, 2017 Enrollment) (Experimental): Group four delayed intervention participants in CO-CSA plus nutrition education will receive a subsidized share of CSA produce (50% standard member price) weekly for approximately 20 weeks in 2018 and will attend nine skill-based, nutrition education sessions focused on use of CSA produce.
  Interventions: Behavioral: CO-CSA plus Nutrition Education

INTERVENTIONS:
Behavioral: CO-CSA plus Nutrition Education — Participants will receive subsidized share of CSA produce (50% standard member price) weekly for approximately 20 weeks each year. In addition, they will attend nine skill-based, nutrition education sessions focused on use of CSA produce.

SUMMARY:
The purpose of this study is to better understand how participation in cost-subsidized community supported agriculture programs paired with tailored education can affect diet quality and energy balance among children in low-income households.

DETAILED DESCRIPTION:
Community Supported Agriculture (CSA) is an innovative approach to increasing consumer access to and consumption of fresh produce, thereby lowering obesity prevalence. However, CSA "share" costs may be a barrier for low-income households with children. This multistate study examines whether subsidizing the cost of CSAs, integrated with tailored education: 1) increases consumption of fruits and vegetables, 2) substitutes fruits and vegetables for more energy-dense foods, and 3) improves overall diet quality and energy balance, thus helping children maintain healthy body weights. It also investigates how cost-offset CSAs ("CO-CSAs") contribute to local agricultural economies. Given the well-documented risk for obesity and limited access to fresh produce among low-income individuals, those households are the target of the intervention in four geographically-diverse states: Vermont, New York, North Carolina and Washington.

FORMATIVE AND LONGITUDINAL RESEARCH: Qualitative and quantitative research is being used to inform implementation of the randomized trial, refine outcome assessment strategies, and provide information needed to design a tailored curriculum to enhance low-income households' knowledge, skills, attitudes, and behaviors related to the use of CSA produce and healthy eating.

In the first year of the study, the investigators conducted interviews and focus groups with stakeholders to gather in-depth data related to the potential of CO-CSA operations to meet the needs and preferences of low-income households and the types of information that would be most valuable to include in the study's curriculum. Key stakeholder groups included adults and children from low-income households, CSA farmers, current full-paying CSA members, and nutrition educators.

The investigators also are conducting a longitudinal quantitative examination of dietary behaviors among current CO-CSA participants in an existing statewide program in Vermont. Using online surveys, the investigators are measuring dietary outcomes quarterly among children, and biannually among adults, from low-income households in the program. Data from Year 1 was used to inform the intervention, while data from subsequent time points will provide an opportunity for analysis of longitudinal patterns.

RANDOMIZED INTERVENTION: In the second phase of the project, the investigators will implement and evaluate a three-year delayed intervention randomized controlled trial of CO-CSA plus skill-based, CSA-tailored education in the four states. The investigators will compare changes in dietary behaviors, reported consumption, energy intake, and weight status parameters between children aged 2-12 in 120 control and 120 intervention households. Two hundred households were enrolled in 2016 and an additional 40 households will be enrolled in 2017. Participant households enrolled in 2016 will receive a CO-CSA share for two seasons and education during their first CO-CSA season (Y1 for intervention households and Y2 for control households). Households enrolled in 2017 will receive a CO-CSA share and education for one season (Y2 for intervention households and Y3 for control households). In addition to outcomes with participants, investigators will conduct economic analysis to evaluate the impact of CO-CSA for farms and communities. While these analyses are not related to the human participants, they are central to the overall project goals.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking
* Parent or legal guardian of a child in the household between the ages of two and 12 years
* Self-reported income less than 185% of the Federal Poverty Level or report enrollment in SNAP, WIC, or Head Start
* Has access to a computer from which s/he can complete on-line data collection
* Has an active e-mail account or willing to create an e-mail account
* Has not participated in CSA in the past three years
* Willing to purchase the 50% CO-CSA share (can use SNAP benefits if desired and available)
* Willing to attend CSA-tailored education sessions
* Willing to make a firm commitment to three years of participation (2016 enrollment) or two years of participation (2017 enrollment), with timing of the off-set benefit determined by randomization
* Complete baseline survey
* Pay deposit to farm

Exclusion Criteria:

* Non-English-speaking
* Not the parent or legal guardian of a child in the household between the ages of two and 12 years
* Self-reported income equal to or greater than 185% of the Federal Poverty Level and no report of SNAP, WIC, or Head Start enrollment
* Does not have access to a computer from which s/he can complete on-line data collection
* Does not have an active e-mail account or is not able or willing to create an e-mail account
* Has participated in CSA in the past three years
* Not able or willing to purchase the 50% CO-CSA share
* Not able or willing to attend CSA-tailored education sessions
* Not able or willing to make a firm commitment to three years of participation (for 2016 enrollment) or two years of participation (2017 enrollment), with timing of the off-set benefit determined by randomization
* Not able or willing to complete baseline survey
* Not able or willing to pay deposit to farm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 305 (Actual)
Dates: Start 2015-04; Primary Completion 2018-12-06 (Actual); Study Completion 2021-03-14 (Actual)

PRIMARY OUTCOMES:
Change in child's fruit and vegetable intake as measured by short dietary screener | Baseline to 4 months, 12 month follow-up, 16-month follow-up, 24-month follow-up, and 28-month follow-up
  Data collected using the National Cancer Institute's All-Day Fruit and Vegetable Screener.
Change in child's fruit and vegetable intake as measured by 24-hour dietary recall | Baseline to 4 months, 16-month follow-up, and 28-month follow-up
  Data collected with dietary recalls using the online Automated Self-Administered 24-Hour Dietary Recall (ASA24) system
Change in child's intake of sugar-sweetened beverages and processed snacks as measured by short dietary questionnaire | Baseline to 4 months, 12-month follow-up, 16-month follow-up, 24-month follow-up, and 28-month follow-up
  Data collected using the Fred Hutchison Cancer Research Center's 'Beverage and Snack Questionnaire 2'
Change in child's intake of sugar-sweetened beverages and processed snacks as measured by 24-hour dietary recall | Baseline to 4 months, 16-month follow-up, and 28-month follow-up
  Data collected with dietary recalls using the online Automated Self-Administered 24-Hour Dietary Recall (ASA24) system
Change in child's caloric intake as a percent of estimated energy requirements | Baseline to 4 months, 16-month follow-up, and 28-month follow-up
  Data collected with dietary recalls using the online Automated Self-Administered 24-Hour Dietary Recall (ASA24) system
Change in child's dermal carotenoid levels | Baseline to 4 months, 16-month follow-up, and 28-month follow-up
  Carotenoid levels measured by resonance Raman spectroscopy using the Bio-Photonic Scanner (NuSkin Enterprises)
Change in child's diet quality | Baseline to 4 months, 16-month follow-up, and 28-month follow-up
  Data collected with dietary recalls using the online Automated Self-Administered 24-Hour Dietary Recall (ASA24) system

SECONDARY OUTCOMES:
Change in child's BMI percentile | Baseline to 4 months, 16-month follow-up, and 28-month follow-up
  Height and weight measured by trained research staff
Change in child's physical activity | Baseline to 4 months, 12 month follow-up, 16-month follow-up, 24-month follow-up, and 28-month follow-up
  Data collected using survey question on physical activity adapted from Youth Risk Behavior Surveillance System (YRBSS) questionnaire
Change in child's sedentary behavior | Baseline to 4 months, 12 month follow-up, 16-month follow-up, 24-month follow-up, and 28-month follow-up
  Data collected using survey questions on TV, video, and computer use adapted from Youth Risk Behavior Surveillance System (YRBSS) questionnaire
Changes in parent's ability to select, store, and prepare CSA produce | Baseline to 4 months, 16-month follow-up, and 28-month follow-up
  Data collected using questionnaire module on parent's ability to select, store, and prepare CSA produce
Changes in parent's ability to prepare foods to minimize added (solid) fat and sugar | Baseline to 4 months, 16-month follow-up, and 28-month follow-up
  Data collected using questionnaire module on parent's ability to prepare foods to minimize added (solid) fat and sugar
Changes in parent's ability to substitute fruit and vegetables for energy-dense foods | Baseline to 4 months, 16-month follow-up, and 28-month follow-up
  Data collected using questionnaire module on parent's ability to substitute fruit and vegetables for energy-dense foods
Changes in parent's knowledge, attitudes, and beliefs about fruits and vegetables | Baseline to 4 months, 16-month follow-up, and 28-month follow-up
  Data collected using questionnaire module on parent's knowledge, attitudes, and beliefs about fruits and vegetables
Changes in availability and accessibility of fruits and vegetables in the home | Baseline to 4 months, 16-month follow-up, and 28-month follow-up
  Data collected using questionnaire module on the availability and accessibility of fruits and vegetables in the home
Change in parent's fruit and vegetable intake as measured by short dietary screener | Baseline to 4 months, 12 month follow-up, 16-month follow-up, 24-month follow-up, and 28-month follow-up
  Data collected using the National Cancer Institute's All-Day Fruit and Vegetable Screener
Change in parent's intake of sugar-sweetened beverages and processed snacks as measured by short dietary questionnaire | Baseline to 4 months, 12 month follow-up, 16-month follow-up, 24-month follow-up, and 28-month follow-up
  Data collected using the Fred Hutchison Cancer Research Center's 'Beverage and Snack Questionnaire 2'
Change in parent's dermal carotenoid levels | Baseline to 4 months, 16-month follow-up, and 28-month follow-up
  Carotenoid levels measured by resonance Raman spectroscopy using the Bio-Photonic Scanner (NuSkin Enterprises)
Changes in household food security | Baseline to 4 months, 12 month follow-up, 16-month follow-up, 24-month follow-up, and 28-month follow-up
  Data collected using the USDA 6-item Food Security Survey Module with 30-day reference period

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca A. Seguin, PhD, Principal Investigator — Cornell University; Karla Hanson, PhD, Principal Investigator — Cornell University; Jane Kolodinsky, PhD, Principal Investigator — University of Vermont; Marilyn Sitaker, PhD, Principal Investigator — The Evergreen State College; Alice Ammerman, PhD, Principal Investigator — University of North Carolina, Chapel Hill; Stephanie Jilcott-Pitts, PhD, Principal Investigator — East Carolina University
Locations (25):
- United States (25):
  - Barker, Barker, New York
  - Corning, Corning, New York
  - Gasport, Gasport, New York
  - Lockport, Lockport, New York
  - Medina, Medina, New York
  - Newfane, Newfane, New York
  - Watertown, Watertown, New York
  - Chapel Hill, Chapel Hill, North Carolina
  - Pittsboro, Pittsboro, North Carolina
  - Siler City, Siler City, North Carolina
  - Bristol, Bristol, Vermont
  - Burlington, Burlington, Vermont
  - Cuttingsville, Cuttingsville, Vermont
  - Hinesburg, Hinesburg, Vermont
  - Ludlow, Ludlow, Vermont
  - Rutland, Rutland, Vermont
  - South Burlington, South Burlington, Vermont
  - Starksboro, Starksboro, Vermont
  - Vergennes, Vergennes, Vermont
  - Winooski, Winooski, Vermont
  - La Conner, La Conner, Washington
  - Mount Vernon, Mount Vernon, Washington
  - Olympia, Olympia, Washington
  - Rochester, Rochester, Washington
  - Sedro Woolley, Sedro-Woolley, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Garner JA, Hanson KL, Jilcott Pitts SB, Kolodinsky J, Sitaker MH, Ammerman AS, Kenkel D, Seguin-Fowler RA. Cost analysis and cost effectiveness of a subsidized community supported agriculture intervention for low-income families. Int J Behav Nutr Phys Act. 2023 Jul 10;20(1):84. doi: 10.1186/s12966-023-01481-7. PMID 37430305
- [Derived] Seguin-Fowler RA, Hanson KL, Jilcott Pitts SB, Kolodinsky J, Sitaker M, Ammerman AS, Marshall GA, Belarmino EH, Garner JA, Wang W. Community supported agriculture plus nutrition education improves skills, self-efficacy, and eating behaviors among low-income caregivers but not their children: a randomized controlled trial. Int J Behav Nutr Phys Act. 2021 Aug 31;18(1):112. doi: 10.1186/s12966-021-01168-x. PMID 34461931
- [Derived] Lu I, Hanson KL, Jilcott Pitts SB, Kolodinsky J, Ammerman AS, Sitaker M, Wang W, Volpe LC, Belarmino EH, Garner J, Gonsalves L, Seguin RA. Perceptions of nutrition education classes offered in conjunction with a community-supported agriculture intervention among low-income families. Public Health Nutr. 2021 Jul;24(10):3028-3036. doi: 10.1017/S1368980020002773. Epub 2020 Aug 24. PMID 32830626
- [Derived] Seguin RA, Morgan EH, Hanson KL, Ammerman AS, Jilcott Pitts SB, Kolodinsky J, Sitaker M, Becot FA, Connor LM, Garner JA, McGuirt JT. Farm Fresh Foods for Healthy Kids (F3HK): An innovative community supported agriculture intervention to prevent childhood obesity in low-income families and strengthen local agricultural economies. BMC Public Health. 2017 Apr 8;17(1):306. doi: 10.1186/s12889-017-4202-2. PMID 28390403